CLINICAL TRIAL: NCT03544866
Title: The Impact of Pediatric Skin Disorders: The "Big" Study
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Pediatric Dermatology Research Alliancce (Unknown); Regeneron Pharmaceuticals (Industry); Immunex Corporation (Industry)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Other Study IDs: ASP02172016
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pediatric Skin Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study leverages the availability of a validated series of instruments to measure the effect of highly visible, chronic skin disorders, including atopic dermatitis (AD), on patients 8 years of age and above in causing stigma and psychiatric issues, particularly anxiety and depression.

DETAILED DESCRIPTION:
This is a multi center study with Northwestern University/Lurie Children's Hospital serving as the Data Coordinating Center. Site selection has been completed through members of PeDRA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be aged 8-17 years of age
* Subject must be diagnosed with a chronic skin disease deemed to be severe enough and/or in a visible location that could be stigmatizing as determined by the study doctor
* Subject and parent must both be English speaking with at least one parent/guardian who will complete the questionnaires
* Subject and Parent/Guardian must be able to complete the relevant questionnaires

Exclusion Criteria:

* Children under 8 years of age
* Children with developmental delay and/or a behavioral disorder that would preclude participation in form completion
* Children with a non-cutaneous disorder that is considered by the Study doctor to be stigmatizing

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 3,500 parent/child dyads across all sites (at least 50 parent/child dyads at each site).
Sampling Method: Non-Probability Sample
Enrollment: 1666 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Measure the stigma experienced by children as a function of the child's perceived skin lesion visibility using the altered Neuro-QoL stigma tool | Past 7 days
  Measure the stigma experienced by children as a function of the child's perceived skin lesion visibility using the altered Neuro-QoL stigma tool

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, Principal Investigator — Northwestern University
Locations (1):
- Department of Dermatology, Northwestern University Feinberg School of Medicine and Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No